CLINICAL TRIAL: NCT02487056
Title: A Multicentre, Prospective, Observational, Hospital-based Registry of Patients With Acute Heart Failure Those Whose Care Was Guided by a Cardiologist in Turkey
Brief Title: Patient Journey in Hospital With Heart Failure in Turkish Population
Acronym: JournayHF-TR
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Mehdi Zoghi, Prof. Dr., Ege University
Other Study IDs: JournayHF-TR
Record Dates: First submitted 2015-06-23; First posted 2015-07-01 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: Heart Failure; Diagnosis; Management
MeSH Terms: conditions — Heart Failure; Disease | interventions — Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized AHF: Patients who were hospitalized with a diagnosis of AHF in the intensive care unit (ICU)/coronary care unit and cardiology wards
  Interventions: Behavioral: Demographic and clinical characteristics, clinical history, symptoms and signs, initial emergency department evaluation, and subsequent inpatient management of HF patients

INTERVENTIONS:
Behavioral: Demographic and clinical characteristics, clinical history, symptoms and signs, initial emergency department evaluation, and subsequent inpatient management of HF patients — Demographic and clinical characteristics, clinical history, symptoms and signs, initial emergency department evaluation, and subsequent inpatient management of patients were recorded.

SUMMARY:
The purpose of this study is to compose a national database of the etiologies, clinical and demographic characteristics, using diagnostic tests, precipitating and risk factors, management of from intensive care unit or coronary care unit to hospital discharge, length of stay in the intensive care unit and hospital, in-hospital mortality and discharge medications of hospitalized acute heart failure patients in Turkish population.

DETAILED DESCRIPTION:
The etiologies, precipitating factors, demographics, clinical characteristics, management and outcome of patients admitted in hospital with acute heart failure in Turkish population will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years olds
* Clinical diagnosis of acute heart failure
* Admitted to the participating hospitals

Exclusion Criteria:

* Patients <18 years old
* Patients with acute heart failure who are discharged from the emergency room without admission.
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with acute heart failure
Sampling Method: Probability Sample
Enrollment: 1622 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Ekmekçi, MD, Study Chair — Dr. Siyami Ersek Göğüs Kalp Ve Damar Cerrahisi Eğitim Ve Araştırma Hastanesi
Locations (1):
- Ahmet Ekmekçi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sinan UY, Ekmekci A, Ozbay B, Akyildiz Akcay F, Bekar L, Koza Y, Bolat I, Kocabas U, Zoghi M; Collaborators. The real-life data of hospitalized patients with heart failure: On behalf of the Journey HF-TR study investigators. Anatol J Cardiol. 2019 Jan;21(1):25-30. doi: 10.14744/AnatolJCardiol.2018.50880. PMID 30587703
- [Result] Sabanoglu C, Sinan UY, Akboga MK, Coner A, Gok G, Kocabas U, Bekar L, Gazi E, Cengiz M, Kilic S, Inanc IH, Cakmak HA, Zoghi M. Long-Term Prognosis of Patients with Heart Failure: Follow-Up Results of Journey HF-TR Study Population. Anatol J Cardiol. 2023 Jan;27(1):26-33. doi: 10.14744/AnatolJCardiol.2022.2171. PMID 36680444

RESULTS

PARTICIPANT FLOW:
Groups:
- JourneyHF-TR: The patients who were hospitalized with the diagnosis of acute heart failure in intensive/coronary care units between September 2015 and 2016 were included in our study.
Period: Overall Study
Arm/Group | JourneyHF-TR
Started | 1622
Completed | 1606
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | JourneyHF-TR
Number analyzed (Participants) | 1606
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 688
  Male | 918

OUTCOME MEASURES:

1. Primary Outcome: Adherence to European Heart Failure Guideline
Description: To assess number of patients managed and treated following the last European Heart Failure Guidelines
Time Frame: Admission to Hospital (Enrollment)
Measure: Count of Participants; unit: Participants
Groups:
- Hospitalized Patients With Acute Heart Failure: The patients who were hospitalized with the diagnosis of acute heart failure in intensive/coronary care units
Arm/Group | Hospitalized Patients With Acute Heart Failure
Number analyzed (Participants) | 1606
Participants | 1172

2. Secondary Outcome: Length of Hospitalisation
Description: Length of stay in hospital in Turkish population admitted to study
Time Frame: In-Hospital
Measure: Median (Full Range); unit: Day
Arm/Group | JourneyHF-TR
Number analyzed (Participants) | 1606
Day | 3 [1 to 72]

3. Secondary Outcome: Mortality
Description: All cause death
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | JourneyHF-TR
Number analyzed (Participants) | 1606
Participants | 122

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Hospitalized Patients With Acute Heart Failure: The Journey HF-TR study is a cross-sectional, multicenter, non-invasive and observational trial that was conducted in intensive/coronary care units and cardiology wards. The patients who were hospitalized with the diagnosis of acute heart failure in intensive/coronary care units between September 2015 and 2016 were included in our study.
Arm/Group | Hospitalized Patients With Acute Heart Failure
All-Cause Mortality (participants affected / at risk) | 122/1606
Serious Adverse Events (participants affected / at risk) | 0/1606
Other Adverse Events (participants affected / at risk) | 0/1606

LIMITATIONS AND CAVEATS:
Although participant sites were encouraged to enroll patients, as consecutively as possible, the study population may not represent the general population. Registry data are based only on documentation of medical history and management during hospitalization, and follow-up data are not obtained. The medication dosage was not recorded, so we are not sure if the patients are taking the appropriate doses of HF medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes